CLINICAL TRIAL: NCT02848547
Title: The Role of Information Technology in the Prevention of Type 2 Diabetes - An Extended Follow-up Study
Brief Title: Post Trial Analysis of a Primary Prevention Study in Asian Indians
Status: Completed | Type: Observational
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: IDRFARH010
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and blood cells are stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention - SMS: Participants in the intervention group received periodic text messages on healthy lifestyle throughout the study period.
  Interventions: Behavioral: Text Messaging via Short Message Service
- Control - Standard Care: Participants in the control group received standard one time advice at entry in the study.

INTERVENTIONS:
Behavioral: Text Messaging via Short Message Service
  Groups: Intervention - SMS

SUMMARY:
An extended follow-up study of NCT00819455 conducted 5 years post randomization. In this study we estimate the incidence of type 2 diabetes among participants enrolled in the diabetes prevention programme. This will provide comparison of the progression to diabetes among group motivated through text messages and the group educated only during enrollment. A total of 537 participants were enrolled in the primary study and are invited to participate in a follow-up visit 3 years post active trial period.

ELIGIBILITY:
Inclusion Criteria:

Participants of the primary prevention programme - NCT00819455.

Exclusion Criteria:

Unwilling for participation

Ages: 40 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants randomized (n=537) in the primary study NCT00819455.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes among participants enrolled in the diabetes prevention programme. | Two years

SECONDARY OUTCOMES:
Long-term impact of healthy lifestyle through mobile phone based text messaging | Two years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nanditha A, Snehalatha C, Raghavan A, Vinitha R, Satheesh K, Susairaj P, Simon M, Selvam S, Ram J, Naveen Kumar AP, Godsland IF, Oliver N, Johnston DG, Ramachandran A. The post-trial analysis of the Indian SMS diabetes prevention study shows persistent beneficial effects of lifestyle intervention. Diabetes Res Clin Pract. 2018 Aug;142:213-221. doi: 10.1016/j.diabres.2018.05.042. Epub 2018 May 31. PMID 29859274